CLINICAL TRIAL: NCT00242788
Title: A Phase I/II, Multicentre Clinical Study Of ZD1839 (Iressa™) In Combination With Capecitabine (Xeloda™) In Subjects With Advanced Colorectal Carcinoma After Failure Of First-Line Chemotherapy
Brief Title: IRESSA™ In Combo With Xeloda™ in Advanced Colorectal Cancer Patients After 1st-Line Chemo Failure
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1839IL/0505
Record Dates: First submitted 2005-10-20; First posted 2005-10-21 (Estimated); Last update posted 2009-04-23 (Estimated); Status verified 2009-04

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Gefitinib; Capecitabine

INTERVENTIONS:
Drug: Gefitinib and capecitabine

SUMMARY:
The primary objective of the Phase I part of the study is to determine the recommended dose of capecitabine to be administered in combination with ZD1839 250 mg orally once daily in subjects with advanced or metastatic colorectal cancer by assessing DLTs.

The primary objective of the Phase II part of the study is to estimate the objective response rate (complete response [CR] and partial response [PR]) at study closure for ZD1839 administered in combination with capecitabine in subjects with advanced or metastatic colorectal cancer using the Response Evaluation Criteria in Solid Tumours (RECIST).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older, Histologically-confirmed colorectal carcinoma, Non-resectable metastatic or locally advanced disease, Objective progression after one prior chemotherapeutic regimen for metastatic or locally advanced disease with an interval of at least 4 weeks between the last administration of chemotherapy and the first administration of study treatment, Measurable lesion according to the RECIST, life expectancy more than 12 weeks, World Health Organisation (WHO) performance status of 0, 1 or 2.

Exclusion Criteria:

* 1. Prior adjuvant chemotherapy if the disease-free interval is less than 6 months Known leptomeningeal or central nervous system (CNS) metastases Known severe hypersensitivity to ZD1839 or any of the excipients of this product Known, severe hypersensitivity to capecitabine or any of the excipients of this product Any evidence of clinically active interstitial lung disease (subjects with chronic stable radiographic changes who are asymptomatic need not be excluded) Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of basal cell carcinoma or cervical cancer in situ Any unresolved chronic toxicity greater than CTC grade 1 from previous anticancer therapy Absolute neutrophil count (ANC) less than 1500 mm3 (1.5 x 109/litre [L]), platelets less than 100 000 mm3 (100 x 109/L) or haemoglobin less than 10 g/dl Serum bilirubin greater than 1.5 times the upper limit of the reference range (ULRR) Serum creatinine greater than 1.25 times the ULRR Creatinine clearance below 30 mL/min (Cockroft and Gault) Alkaline phosphatase (ALP) greater than 5 times the ULRR or greater than 20 times the ULRR in subjects with known bone metastasesAlanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than 2.5 times the ULRR if no demonstrable liver metastases, or greater than 5 times the ULRR in the presence of liver metastases Prothrombin time (PT) or activated partial thromboplastin time (aPTT) less than 70% normal laboratory value As judged by the investigator, any evidence of severe or uncontrolled systemic disease (e.g., unstable or uncompensated respiratory, cardiac, hepatic, or renal disease) Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the subject to participate in the study Pregnancy or breast feeding (women of child-bearing potential) Concomitant use of phenytoin, carbamazepine, rifampicin or barbiturates Treatment with a non-approved or investigational drug within 30 days before Day 1 of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-02; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Objective tumour response (CR and PR) at study closure based on the RECIST

SECONDARY OUTCOMES:
Incidence of controlled disease (CR, PR and SD) at study closure

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Spain Medical Director, MD, Study Director — AstraZeneca
Locations (6):
- Spain (6):
  - Research Site, Girona
  - Research Site, Leganés
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Santander
  - Research Site, Zaragoza